CLINICAL TRIAL: NCT06103838
Title: A Phase II Trial Evaluating 18F-Fluciclovine PET/CT in Multiple Myeloma
Brief Title: 18F-Fluciclovine PET/CT in Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001525; 001525-C
Record Dates: First submitted 2023-10-26; First posted 2023-10-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-08-18

CONDITIONS: Multiple Myeloma; Newly Diagnosed Multiple Myeloma (NDMM); Relapsed and/or Refractory Multiple Myeloma (RRMM)
Keywords: RRMM; NDMM; 18F-FDG PET/CT; PET/CT; 18F-fluciclovine; Imaging; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-fluciclovine PET/CT in Multiple Myeloma (Experimental): Evaluate 18F-fluciclovine PET/CT in participants with multiple myeloma at Timepoint #1, Timepoint #2 ( after induction treatment (NDMM) or six months (RRMM)) and at Timepoint #3 (the time of progression or 5 years).
  Interventions: Drug: 18F-fluciclovine injection; Procedure: 18F-FDG PET/CT

INTERVENTIONS:
Drug: 18F-fluciclovine injection — 370 MBq (10 mCi)(+/-20%) as a bolus intravenous injection.
Procedure: 18F-FDG PET/CT — All participants will undergo 18F-FDG PET/CT within 30 days of the 18F-fluciclovine PET/CT scan

SUMMARY:
Background:

Multiple myeloma (MM) is an incurable cancer of certain blood cells. MM often returns after treatment, and most people survive only 5 to 8 years after diagnosis. To improve survival, researchers need to find ways to identify returning disease earlier.

Objective:

To find out if the radiotracer 18F-fluciclovine (a substance injected into the blood during imaging scans) is better at detecting MM than the one (18F-FDG) currently used for this purpose.

Eligibility:

Adults aged 18 years or older with MM. The MM may be newly diagnosed (NDMM); or it may have returned or failed to respond after at least 1 prior line of treatment (RRMM).

Design:

Participants will be screened. They will have blood tests. They will have a positron emission tomography (PET) or computed tomography (CT) scan using 18F-FDG. The radiotracer will be injected into a vein. Then participants will lie on a table while the PET/CT scan takes images of their body.

All participants will have 3 study visits. During each visit they will have:

Two PET/CT scans. One with 18F-FDG, one with 18F-fluciclovine.

An optional magnetic resonance imaging scan.

A bone marrow biopsy. An area on the hip will be numbed; a needle will be inserted to draw out a sample of the soft tissue from inside the bone.

These tests may be spread over 30 days for each visit.

NDMM participants will have their second study visit 2 to 4 weeks after they complete their usual treatment for the disease. RRMM participants will have their second visit 6 months after their first.

All participants will have a third study visit after 5 years or when their disease progresses.

DETAILED DESCRIPTION:
Background:

* Multiple myeloma (MM) is an incurable malignancy of plasma cells that leads to destructive bone lesions, renal damage, anemia, and hypercalcemia. MM is the second most common hematologic malignancy. The American Cancer Society estimates that annually over 34,000 new cases of MM will occur in the U.S. and over 12,000 deaths due to MM in 2022.
* Overall survival (OS) has improved significantly over the past 20 years with the development of proteasome inhibitors (PIs), immunomodulatory agents (IMiDs) and anti-CD38 monoclonal antibodies. However, despite these advances, patients ultimately relapse requiring multiple subsequent lines of therapy. As MM evolves, it generally becomes more refractory, and patients ultimately succumb to their disease.
* With multiple lines of efficacious therapies, the correct early identification of relapsed disease is important to trigger initiation of a new line of therapy.
* Limitations in conventional imaging highlight a need for molecular imaging agents with better sensitivity for detecting and measuring tumor burden to improve staging and treatment selection for patients with MM and plasma cell dyscrasias.
* 18F-fluciclovine is a radionuclide approved by the FDA for evaluating suspected prostate cancer recurrence but has shown additional ability in detecting MM lesions.

Objective:

To determine the concordance between 18F-fluciclovine PET/CT and 18F-FDG PET/CT in participants with multiple myeloma

Eligibility:

* Participants >= 18 years old
* Eastern Cooperative Oncology Group (ECOG) Performance score of 0 to 2
* Participants must have a documented diagnosis of MM defined by the International Myeloma Working Group (IMWG) Criteria
* Participants fit criteria for one of the following categories:

  * Newly diagnosed multiple myeloma (NDMM) without previous treatment (or within the first 3 cycles of front-line treatment)
  * Relapsed and/or Refractory multiple myeloma (RRMM) with at least 1 prior line of therapy

Design:

This is an open-label, single center phase 2 study evaluating 18F-fluciclovine PET/CT imaging in up to 50 participants with multiple myeloma. Participants will be enrolled into one of two cohorts based on disease status; newly diagnosed multiple myeloma (NDMM) participants will be enrolled into Cohort 1 and relapsed refractory multiple myeloma (RRMM) participants will be enrolled into Cohort 2. All subjects will undergo an 18F-fluciclovine injection followed by a static whole-body PET/CT at three time points: Timepoint #1, Timepoint #2 (after induction for NDMM or at 6 months for RRMM) and Timepoint #3 (at progression or at 5 years). Results will be compared to 18F-FDG PET/CT imaging at those same timepoints.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have a documented diagnosis of MM defined by the IMWG Criteria. Participants at diagnosis must have had a serum M-protein >= 3 g/dL and/or bone marrow plasma cells >= 10% and at least one of the following:

  * Anemia: Hemoglobin <=10 g/dL, or
  * Renal Failure: serum creatinine >= 2.0 mg/dL, or
  * Hypercalcemia: Ca >= 10.5 mg/dL, or
  * Lytic bone lesions on X-ray, CT, or PET/CT, or
  * >= 2 focal lesions on spinal MRI, or
  * >= 60% bone marrow plasma cells, or
  * Involved/un-involved serum free light chain ration >= 100
* Participants must have measurable disease defined by any one of the following:

  * Monoclonal bone marrow plasma cells > 5%
  * Serum monoclonal protein >= 0.2 g/dl
  * Urine monoclonal protein > 200 mg/24 hr
  * Serum immunoglobulin free light chain > 10 mg/dL AND abnormal kappa/lambda ratio
  * A measurable lesion on PET/CT or MRI
* Participants fit criteria for one of the following categories:

  * Newly diagnosed multiple myeloma (NDMM)
  * Relapsed and/or refractory multiple myeloma (RRMM) with at least 1 prior line of therapy
* Age >=18 years.
* ECOG performance status <= 2
* Negative serum or urine pregnancy test at screening for WOCBP.
* Women of child-bearing potential and men must agree to use effective contraception (hormonal or barrier method of birth control; abstinence) 24 hours prior to and for the 24 hours after each 18F-fluciclovine administration.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 18F-FDG
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 18F-fluciclovine or other similar agents.
* Subjects with severe claustrophobia unresponsive to oral anxiolytics or unwilling to take them.
* Uncontrolled intercurrent illness including, psychiatric illness/social situations that would limit compliance with study requirements.
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 18F-fluciclovine, breastfeeding should be discontinued if the mother is treated with 18F-fluciclovine until 3 days after 18F-fluciclovine.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-12-06 (Estimated); Study Completion 2031-12-06 (Estimated)

PRIMARY OUTCOMES:
To determine the concordance between 18F-fluciclovine PET/CT and 18F-FDG PET/CT in participants with multiple myeloma. | After 50 evaluable participants have completed baseline scans.
  The performance of 18F-fluciclovine PET/CT is assessed by concordance with the 18F-FDG PET/CT imaging in scan positivity. A positive lesion is defined as focal uptake greater than background associated with abnormal CT findings (i.e., lytic bone lesions or extramedullary tissue.) The point estimates and 95% confidence intervals of the concordance rate in scan positivity between 18F-fluciclovine and 18F-FDG PET/CT will be reported.

SECONDARY OUTCOMES:
Evaluate the efficacy of 18F-fluciclovine in measuring disease volume as compared to other indicators of disease volume such as serum M protein, serum free-light chains, urine M protein, B2 microglobulin, and bone marrow plasma cell percentage. | Between Timepoint #1 and Timepoint #3
  Disease volumes measured by 18F-fluciclovine will be correlated with other indicators of disease volume such as serum M protein, serum free-light chains, urine M protein, B2 microglobulin, and bone marrow plasma cell percentage by Spearman rank correlation.
Evaluate the ability of 18F-fluciclovine to identify minimal residual disease (MRD) as compared to MRD status determined by bone marrow flow cytometry or next generation sequencing (NGS). | Between Timepoint #1 and Timepoint #3
  Status of minimal residual disease (MRD) identified by 18F-fluciclovine will be compared to MRD status determined by bone marrow flow cytometry or next generation sequencing (NGS).
Evaluate the ability for 18F-fluciclovine to evaluate response after treatment as compared to the IMWG response criteria. | Between Timepoint #1 and Timepoint #3
  Response after treatment determined by 18F-fluciclovine will be compared to the IMWG response criteria by McNemar test.
Evaluate the safety of 18F-fluciclovine as a radiotracer in patients with multiple myeloma. | From the time at each 18F-fluciclovine dose through 3 days after each dose.
  All participants will be evaluable for toxicity from the time at each 18F-fluciclovine dose through 3 days after each dose. Safety of the agents will be assessed by determining the type, grade, and frequency of adverse events noted in each participant who receives at least one dose of each of the study treatments. Safety data will be presented in a summary.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Hill, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be made available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available upon request and with the permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001525-C.html